CLINICAL TRIAL: NCT00797914
Title: Phase I Study for Evaluation of Handheld Colonoscopy Force Monitor by Expert Endoscopists in the Performance of Colonoscopy
Brief Title: Evaluation of Handheld Colonoscopy Force Monitor by Expert Endoscopists in the Performance of Colonoscopy
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Capital Digestive Care, LLC (Other); Mayo Clinic (Other); Sansum Clinic (Unknown); Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: CFM-01; 5R44DK068936 (NIH)
Record Dates: First submitted 2008-11-23; First posted 2008-11-25 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Identify Characteristics of Colonoscopists During Endoscopy
Keywords: Colonoscopy; Instrumentation; Force Monitoring; Quality Control; Training

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing colonoscopy: Patients who are undergoing outpatient colonoscopy for colorectal cancer screening or for symptoms suggestive of colonic diseases.

SUMMARY:
The purpose of this study is to evaluate a handheld Colonoscopy Force Monitor(CFM™), a push-pull force and torque measuring device, that grips the shaft of the colonoscope and wirelessly transmits and records all the forces applied by the endoscopist during colonoscopy.

DETAILED DESCRIPTION:
Colonoscopy requires a skilled endoscopist to use visual and tactile information to advance and withdraw the instrument through a series of fixed and stationary loops. To develop and maintain the skills necessary to perform colonoscopy safely and effectively requires extensive training and ongoing education. Quantification of tactile information provides the opportunity to understand the "feel" used by the endoscopist to perform colonoscopy. The identification of force application patterns has the potential to enhance training and improve performance. CFM™ is a handheld device that uses load cells to transform applied force to electric signals and to transmit wirelessly the signal to a computer for storage and visual display. The device is designed so that the endoscopist maintains a conventional hand position and uses an electronically controlled grip and release mechanism to fix the position on the instrument. Several expert endoscopists from multiple institutions will use the CFM™ to perform colonoscopy. The data will be recorded and analyzed for differences by patient characteristics(e.g. gender, age, pain sensation, surgical history) and by endoscopist.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age: 30-75 years
* ASA Class I or II
* All ethnic and racial groups will be included

Exclusion Criteria:

* Colonic pathology that in the opinion of the endoscopist could interfere with the colonoscopy. Examples include: colonic stricture, poor preparation, obstructing tumor.
* Specific pathology that would limit the extent of examination
* ASA class 3 or greater
* Pregnancy
* Monitored anesthesia using propofol for sedation.
* Vulnerable subjects. Students, nursing home residents, institutionalized patients, and those with psychological or physical incapacity

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult male and female patients between the ages of 30 and 75 presenting to the Chevy Chase Endoscopy Center for screening or diagnostic colonoscopy to be performed by any of the investigators will be considered for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2008-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
CFM can continuously record forces applied to colonoscope by different expert endoscopists during routine outpatient colonoscopy. | 1 year

SECONDARY OUTCOMES:
CFM can characterize differences in force patterns for different patients and different endoscopists | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Louis Y Korman, M.D., Principal Investigator — Capital Digestive Care, LLC
Locations (3):
- United States (3):
  - Sansum Clinic, Santa Barbara, California
  - Chevy Chase Endoscopy Center, Chevy Chase, Maryland
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Result] Korman LY, Egorov V, Tsuryupa S, Corbin B, Anderson M, Sarvazyan N, Sarvazyan A. Characterization of forces applied by endoscopists during colonoscopy by using a wireless colonoscopy force monitor. Gastrointest Endosc. 2010 Feb;71(2):327-34. doi: 10.1016/j.gie.2009.08.029. Epub 2009 Nov 17. PMID 19922923